CLINICAL TRIAL: NCT05363683
Title: Optimizing Movement After Anterior Cruciate Ligament Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0652-21-FB; U54GM115458 (NIH)
Record Dates: First submitted 2022-05-02; First posted 2022-05-06 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-06

CONDITIONS: Anterior Cruciate Ligament Injuries; Knee Osteoarthritis
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Osteoarthritis, Knee | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard care
  Interventions: Procedure: Standard Care
- Experimental (Experimental): Squat biofeedback intervention
  Interventions: Procedure: Squat Biofeedback

INTERVENTIONS:
Procedure: Squat Biofeedback — The intervention group will complete bilateral squats with each limb on a separate portable force plate. They will receive real-time visual feedback on a 32-inch screen during all squats. Biofeedback conditions will be progressed from simplest (ground reaction force only) to most complex (ground reaction force plus center of pressure). This intervention will be included in additional to standard care post-operative physical therapy.
  Arms: Experimental
Procedure: Standard Care — The intervention group will receive standard care post-operative physical therapy.
  Arms: Control

SUMMARY:
Fifty percent of teenagers and young adults who suffer an anterior cruciate ligament (ACL) injury develop knee osteoarthritis (OA) within 15 years. The resulting pain, reduced quality-of-life, and increased risk for co-morbidity lead to substantial healthcare costs, inability to fulfill work and personal responsibilities, and reduced long-term health. Degeneration in articular cartilage, connective tissue that covers the ends of bones in the knee, is the hallmark of early OA development after knee injury. This deterioration can be measured by an imaging biomarker for OA development on quantitative magnetic resonance imaging (MRI). Harmful increases in MRI markers of the knee's articular cartilage occur within months of ACL injury and indicate preventative interventions should begin soon after injury. However, evidence-based interventions to prevent OA do not exist.

This project will challenge the traditional OA paradigm that too much joint loading (e.g. "wear and tear") causes cartilage breakdown. A multi-disciplinary team has developed a novel visual biofeedback paradigm using portable force plates that can increase knee loading during squats within a single session after ACL reconstruction (ACLR). This study will determine the efficacy of the visual biofeedback program initiated two weeks after ACLR by assessing movement biomechanics and MRI changes in cartilage after six months later. Successful completion of this project will establish the first rehabilitation intervention to effectively and optimally load the knee joint early after ACLR, providing the initial steps to prevent OA after ACL injury.

DETAILED DESCRIPTION:
Fifty percent of teenagers and young adults who suffer an anterior cruciate ligament (ACL) injury develop radiographic knee osteoarthritis (OA) within 15 years. The resulting pain, reduced quality-of-life, and increased risk for co-morbidity lead to substantial healthcare costs, inability to fulfill work and personal responsibilities, and reduced long-term health. Degeneration in articular cartilage, connective tissue that covers the ends of bones in the knee, is the hallmark of early OA development after knee injury. This deterioration can be measured by increased T2 and T1rho relaxation time on quantitative magnetic resonance imaging (MRI), an imaging biomarker for OA development. Harmful increases in MRI markers of the knee's articular cartilage occur within months of ACL injury and indicate preventative interventions should begin soon after injury. However, evidence-based interventions to prevent OA do not exist. The investigators have shown that after ACL reconstruction (ACLR), patients exhibit asymmetric movement patterns characterized by up to 62% lower knee joint loading during walking and squatting in the injured limb at two months after ACLR. These knee joint loading patterns remain 40% lower at six months. Emerging evidence suggests knee joint unloading patterns after ACL injury may increase the risk for OA development. Currently, no studies have examined the efficacy of movement-focused interventions during the first months after ACLR, which explains the lack of evidence-based interventions that successfully increase knee loading early after ACLR. This gap presents a barrier to the long-term goal of preventing OA in young, active individuals before irreversible knee degeneration occurs. This project will challenge the traditional OA paradigm that too much joint loading (e.g. "wear and tear") causes cartilage breakdown. The multi-disciplinary team spanning rehabilitation, orthopaedics, radiology and biomechanics has developed a novel visual biofeedback paradigm using portable force plates that can increase knee loading during squats within a single session after ACLR. This data suggest movement is modifiable using visual feedback, but its efficacy beyond a single training session is unknown. This study will determine the efficacy of the visual biofeedback program initiated two weeks after ACLR by assessing movement biomechanics and MRI changes in cartilage microstructure six months later. Successful completion of this project will establish the first rehabilitation intervention to effectively and optimally load the knee joint early after ACLR, providing the initial steps in the team's work to prevent OA after ACL injury.

ELIGIBILITY:
Inclusion Criteria:

* Acute anterior cruciate ligament (ACL) injury in the past 6 months
* ACL reconstruction in the past month or have a planned ACL reconstruction

Exclusion Criteria:

* Previous knee injury or surgery (contralateral knee)
* Body mass index (BMI) over 35 kg/m2
* Concomitant posterior cruciate ligament reconstruction or cartilage procedure that includes extended weight bearing restrictions and/or changes to cartilage structure
* Current or planned pregnancy during study duratuiom

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Wellsandt, DPT, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wellsandt MJ, Weldon N, Werner DM, McManigal ML, Tao MA, Rosenthal MD, Sajja BR, Wichman CS, Baker A, Johnson C, Specht Z, Weaver BA, Knarr B, Nabower C, Wellsandt E. Efficacy of a Squat Visual Biofeedback Program After ACL Reconstruction: Protocol for a Prospective, Parallel, Randomized Controlled Trial. Int J Sports Phys Ther. 2025 Sep 2;20(9):1364-1376. doi: 10.26603/001c.142879. eCollection 2025. PMID 40904719

RESULTS

PARTICIPANT FLOW:
Groups:
- Biofeedback Group: Provided real-time visual feedback on a screen during bilateral squat intervention.
- Control Group: Provided standard verbal instructions during bilateral squat intervention.
Period: Overall Study
Arm/Group | Biofeedback Group | Control Group
Started | 16 | 18
Completed | 15 | 17
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: 1 participant in the control group dropped from the study and did not complete any baseline testing.
Groups:
- Total: Total of all reporting groups
Arm/Group | Biofeedback Group | Control Group | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: 1 participant from the control group dropped from the study and did not complete any baseline test; 1 participant from the squat biofeedback group did not complete the demographics survey during baseline testing.
  Years
    number analyzed (Participants) | 15 | 17 | 32
    (all) | 20.9 (6.6) | 19.3 (4.6) | 20.1 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant from the control group dropped from the study and did not complete any baseline test; 1 participant from the squat biofeedback group did not complete the demographics survey during baseline testing.
  Participants
    number analyzed (Participants) | 15 | 17 | 32
    Female | 10 | 5 | 15
    Male | 5 | 12 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 participant from the control group dropped from the study and did not complete any baseline test; 1 participant from the squat biofeedback group did not complete the demographics survey during baseline testing.
  Participants
    number analyzed (Participants) | 15 | 17 | 32
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 2 | 3
    White | 10 | 8 | 18
    More than one race | 1 | 1 | 2
    Unknown or Not Reported | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 participant from the control group dropped from the study and did not complete any baseline test; 1 participant from the squat biofeedback group did not complete the demographics survey during baseline testing.
  Participants
    number analyzed (Participants) | 15 | 17 | 32
    Hispanic or Latino | 3 | 5 | 8
    Not Hispanic or Latino | 12 | 12 | 24
    Unknown or Not Reported | 0 | 0 | 0
Knee Flexion Moment Impulse at Baseline [Mean (Standard Deviation); unit: Ratio] — Participants completed 3 sets of 5 bilateral bodyweight squats with arms crossed at the chest, with the middle 3 of each set (9 total) averaged and reported. The external knee flexion moment was calculated using an inverse dynamics approach. The interlimb ratio (injured limb / uninjured limb) of the knee flexion moment impulse during descent and ascent of bilateral squatting was analyzed at baseline (pre-intervention). A value of 1 represents symmetric knee flexion moment impulse; a value less than 1 represents a smaller knee flexion moment impulse in the injured compared to uninjured limb. Population: 1 participant from the control group dropped from the study and did not complete any baseline testing.
  Ratio | 0.23 (0.19) | 0.26 (0.16) | 0.25 (0.18)
Vertical Ground Reaction Force Impulse at Baseline [Mean (Standard Deviation); unit: Ratio] — Participants completed 3 sets of 5 bilateral bodyweight squats with arms crossed at the chest, with the middle 3 of each set (9 total) averaged and reported. The vertical ground reaction force was measured. The interlimb ratio (injured limb / uninjured limb) of the vertical ground reaction force during descent and ascent of bilateral squatting was analyzed at baseline (pre-intervention). A value of 1 represents symmetric vertical ground reaction force; a value less than 1 represents a smaller vertical ground reaction force in the injured compared to uninjured limb. Population: 1 participant from the control group dropped from the study and did not complete any baseline testing. 1 participant from the squat biofeedback group dropped after part of baseline testing was completed with no follow-up testing completed; therefore, their data was not used as a covariate in ANCOVA analyses.
  Ratio | 0.72 (0.11) | 0.72 (0.12) | 0.72 (0.11)

OUTCOME MEASURES:

1. Primary Outcome: Knee Flexion Moment Impulse
Description: Participants completed 3 sets of 5 bilateral bodyweight squats with arms crossed at the chest, with the middle 3 of each set (9 total) averaged and reported. The external knee flexion moment was calculated using an inverse dynamics approach. The interlimb ratio (injured limb / uninjured limb) of the knee flexion moment impulse during descent and ascent of bilateral squatting was analyzed at post-intervention. A value of 1 represents symmetric knee flexion moment impulse; a value less than 1 represents a smaller knee flexion moment impulse in the injured compared to uninjured limb.
Time Frame: Immediately post-intervention (within approximately 1 week after completing intervention)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Biofeedback Group | Control Group
Number analyzed (Participants) | 15 | 17
Ratio | 0.54 (0.28) | 0.50 (0.21)
Statistical Analysis 1: Comparison: Biofeedback Group vs Control Group; Test type: Superiority; p = 0.293, ANCOVA

2. Primary Outcome: Cartilage T2 Relaxation Time
Description: Percent change in cartilage T2 relaxation time will be measured by a magnetic resonance imaging (MRI) scan. A positive percent change represents longer (worse) T2 relaxation times at 6 months compared to baseline testing.
Time Frame: Baseline (immediately before intervention, 2-6 weeks after anterior cruciate ligament reconstruction) and 6 months after anterior cruciate ligament reconstruction.
Reporting Status: Not Posted, anticipated posting 2026-01

3. Secondary Outcome: Knee Flexion Moment Impulse
Description: Participants completed 3 sets of 5 bilateral bodyweight squats with arms crossed at the chest, with the middle 3 of each set (9 total) averaged and reported. The external knee flexion moment was calculated using an inverse dynamics approach. The interlimb ratio (injured limb / uninjured limb) of the knee flexion moment impulse during descent and ascent of bilateral squatting was analyzed at 6 months. A value of 1 represents symmetric knee flexion moment impulse; a value less than 1 represents a smaller knee flexion moment impulse in the injured compared to uninjured limb.
Time Frame: 6 months after anterior cruciate ligament reconstruction.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Biofeedback Group | Control Group
Number analyzed (Participants) | 15 | 17
Ratio | 0.66 (0.24) | 0.54 (0.21)
Statistical Analysis 1: Comparison: Biofeedback Group vs Control Group; Test type: Superiority; p = 0.114, ANCOVA

4. Secondary Outcome: Vertical Ground Reaction Force Impulse
Description: Participants completed 3 sets of 5 bilateral bodyweight squats with arms crossed at the chest, with the middle 3 of each set (9 total) averaged and reported. The vertical ground reaction force impulse was calculated. The interlimb ratio (injured limb / uninjured limb) of the vertical ground reaction force impulse during descent and ascent of bilateral squatting was analyzed at post-intervention. A value of 1 represents symmetric vertical ground reaction force impulse; a value less than 1 represents a smaller vertical ground reaction force impulse in the injured compared to uninjured limb.
Time Frame: Immediately post-intervention (approximately 1 week after intervention)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Biofeedback Group | Control Group
Number analyzed (Participants) | 15 | 17
Ratio | 0.91 (0.08) | 0.84 (0.11)
Statistical Analysis 1: Comparison: Biofeedback Group vs Control Group; Test type: Superiority; p = 0.017, ANCOVA

5. Secondary Outcome: Vertical Ground Reaction Force Impulse
Description: Participants completed 3 sets of 5 bilateral bodyweight squats with arms crossed at the chest, with the middle 3 of each set (9 total) averaged and reported. The vertical ground reaction force impulse was calculated. The interlimb ratio (injured limb / uninjured limb) of the vertical ground reaction force impulse during descent and ascent of bilateral squatting was analyzed at 6 months. A value of 1 represents symmetric vertical ground reaction force impulse; a value less than 1 represents a smaller vertical ground reaction force impulse in the injured compared to uninjured limb.
Time Frame: 6 months after anterior cruciate ligament reconstruction.
Measure: Mean (Standard Deviation); unit: N/A (Ratio)
Arm/Group | Biofeedback Group | Control Group
Number analyzed (Participants) | 15 | 17
N/A (Ratio) | 0.95 (0.08) | 0.86 (0.10)
Statistical Analysis 1: Comparison: Biofeedback Group vs Control Group; Test type: Superiority; p = 0.021, ANCOVA

6. Secondary Outcome: Peak Knee Flexion Moment
Description: Participants completed 5 valid trials of walking in each limb. The external knee flexion moment was calculated using an inverse dynamics approach. The interlimb ratio (injured limb / uninjured limb) of the peak knee flexion moment during walking was analyzed at post-intervention. A value of 1 represents symmetric peak knee flexion moment; a value less than 1 represents a smaller peak knee flexion moment in the injured compared to uninjured limb.
Time Frame: Immediately post-intervention (within approximately 1 week after completing intervention)
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Biofeedback Group | Control Group
Number analyzed (Participants) | 15 | 17
Ratio | 0.6 [0.2 to 0.8] | 0.7 [0.4 to 0.8]
Statistical Analysis 1: Comparison: Biofeedback Group vs Control Group; Test type: Superiority; p = 0.936, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Peak Knee Flexion Moment
Description: Participants completed 5 valid trials of walking in each limb. The external knee flexion moment was calculated using an inverse dynamics approach. The interlimb ratio (injured limb / uninjured limb) of the peak knee flexion moment during walking was analyzed at 6 months. A value of 1 represents symmetric peak knee flexion moment; a value less than 1 represents a smaller peak knee flexion moment in the injured compared to uninjured limb.
Time Frame: 6 months after anterior cruciate ligament reconstruction.
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Biofeedback Group | Control Group
Number analyzed (Participants) | 15 | 17
Ratio | 0.7 [0.6 to 0.9] | 0.7 [0.6 to 0.9]
Statistical Analysis 1: Comparison: Biofeedback Group vs Control Group; Test type: Superiority; p = 0.867, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Quadriceps Strength
Description: Participants completed 3 trials of maximal isometric quadriceps strength testing using an isokinetic dynamometer at each limb, with the best trial in each limb used for analysis. The interlimb ratio (injured limb / uninjured limb) of maximum quadriceps strength was analyzed at post-intervention. A value of 1 represents symmetric quadriceps strength; a value less than 1 represents less quadriceps strength in the injured compared to uninjured limb.
Time Frame: Immediately post-intervention (within approximately 1 week after completing intervention)
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Biofeedback Group | Control Group
Number analyzed (Participants) | 15 | 17
Ratio | 0.5 [0.4 to 0.6] | 0.5 [0.5 to 0.6]
Statistical Analysis 1: Comparison: Biofeedback Group vs Control Group; Test type: Superiority; p = 0.370, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Quadriceps Strength
Description: Participants completed 3 trials of maximal isometric quadriceps strength testing using an isokinetic dynamometer at each limb, with the best trial in each limb used for analysis. The interlimb ratio (injured limb / uninjured limb) of maximum quadriceps strength was analyzed at 6 months. A value of 1 represents symmetric quadriceps strength; a value less than 1 represents less quadriceps strength in the injured compared to uninjured limb.
Time Frame: 6 months after anterior cruciate ligament reconstruction.
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Biofeedback Group | Control Group
Number analyzed (Participants) | 15 | 17
Ratio | 0.8 [0.5 to 0.8] | 0.6 [0.6 to 0.7]
Statistical Analysis 1: Comparison: Biofeedback Group vs Control Group; Test type: Superiority; p = 0.379, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From study enrollment until 6 months after anterior cruciate ligament reconstruction. Enrollment was completed either before anterior cruciate ligament reconstruction or within 6 weeks after anterior cruciate ligament reconstruction.
Arm/Group | Biofeedback Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT05363683/Prot_SAP_000.pdf